CLINICAL TRIAL: NCT03022474
Title: Kindergarten-based Intervention for Childhood Obesity in Guangzhou(KICOG)
Acronym: KICOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Xiu Qiu, Healthcare Department Director, Guangzhou Women and Children's Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20121A011070
Record Dates: First submitted 2017-01-13; First posted 2017-01-16 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Childhood Obesity
Keywords: Childhood obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Healthy Lifestyles Intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Healthy Lifestyles Intervention — The program included three major components. The first component consists of live lectures to kindergarten staff about basic nutrition and food concepts that attempted to correct false beliefs. The second component was a health curriculum for children that focused on promoting healthy nutrition habits and a healthy living style. Preschools were required to ensure that children received a health education lesson every two weeks. The third component was aimed at educating parents and consisted of lectures every two months, preschool-home communication every week and child growth monitoring every three months.
  Arms: Intervention group

SUMMARY:
Early life interventions for childhood obesity may provide substantial benefits. Most existing studies aimed at school children have reported limited effectiveness, however few have targeted preschool children. This study aimed to pilot procedures for a multifaceted, culturally appropriate intervention for preschool children and to provide a preliminary assessment of effectiveness of the intervention.

DETAILED DESCRIPTION:
The intervention protocol was developed by an expert group from the National Children Obesity Intervention Team, comprising pediatricians, children healthcare doctors, preschool teachers, and nutritionists, and included three integrated components:

Component 1 - training of kindergarten staff: Before the start of the program, two members of the intervention team (a dietitian and a physician) delivered eight 40-min sessions (twice a week for a month) on dietary management in children and daily food purchasing for school doctors and kitchen staff. During the trial, two health education doctors gave lectures every two months on general knowledge in nutrition to all preschool staff, focusing on the promotion of healthy food and restriction of unhealthy food. To assess the effectiveness of these lectures, we administered a questionnaire on the material covered. We also trained the kitchen staff to use the dietary software to plan menu with balanced nutrition for preschool children.

Component 2 - a curriculum promoting healthy diet and lifestyle: We designed a health education curriculum and associated picture books for the children. Children in the intervention group received a 20-minute health education lesson every week, where they had learning activities and games covering healthy food choice, appropriate portion sizes and eating pace, and reduction of sedentary behaviours. Learning aids such as colourful picture books or cards, food models, nursery rhymes and stories were used. Two elements were introduce to increase children's activity such as lunchtime activity and daily dance at less than 10 minutes during break.

Component 3 - collaboration between families and kindergartens: We organized lectures designed for parents every two months during the intervention period. Topics covered included the cause and harms of childhood obesity, advice on healthy diet (increasing consumption of vegetables and fruits, reducing consumption of meat, snacks, fast foods, and eating out, and avoiding sugary drinks), body mass index (BMI) reference for preschool-age children, and how to use growth curves. We produced a handbook for communication between families and schools, to be handed out to every family weekly, in which children's health behaviours were documented and reviewed by teachers and parents. Finally, parents were notified of their children's anthropometric measurements every three months, so that they could plot and interpret their children's growth curves.

ELIGIBILITY:
Inclusion Criteria:

(i) run by the government (public kindergarten); (ii) located in the central area of the district; (iii) had no less than 100 students; (iv)had no less than two school doctors.

Exclusion Criteria:

* None

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 984 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) change | BMI was measured at baseline and one year after intervention
BMI Z-score change | BMI Z-score was measured and calculated at baseline and one year after intervention

SECONDARY OUTCOMES:
Feasibility and acceptability of the intervention | During intervention
  Qualitatively describe

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, Doctor, Study Director — Guangzhou Women and Children's Medical Center, China

IPD SHARING:
Plan to Share IPD: No